CLINICAL TRIAL: NCT07262580
Title: The Feasibility of an Intervention Targeting Sources of Meaning in Cardiac Rehabilitation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Danish Heart Foundation (Other); Odense Municipality, Denmark (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REC610; Grant no. 2023-12404 (Other Grant/Funding Number: The Danish Heart Foundation)
Record Dates: First submitted 2025-09-24; First posted 2025-12-03 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Heart Disease; Mental Health Outcomes; Rehabilitation
Keywords: cardiac rehabilitation; Heart disease; Sources of Meaning Card Method; Intervention; Individual intervention; Dyadic intervention; Group intervention; Sources of Meaning; Feasibility study; Pre-post design; Intervention adherence; Recruitment rate; Acceptability of interventions; Staff perspectives on acceptability and practicality; Patients and relatives
MeSH Terms: conditions — Heart Diseases; Adherence Interventions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- a) Individual intervention format (Experimental): 1:1 conversation between a professional and a patient in rehabilitation.
  Interventions: Other: Conversation on Sources of Meaning in life with heart disease
- b) Dyadic (patient-relative) intervention format (Experimental): The patient participates together with a relative and a professional.
  Interventions: Other: Dyadic Conversation on Sources of Meaning in Life with heart disease
- c) Group based intervention format (Experimental): A group-based approach, where approximately 6-10 patients in rehabilitation meet for a group session.
  Interventions: Other: Group based session on Sources of Meaning in life with heart disease

INTERVENTIONS:
Other: Conversation on Sources of Meaning in life with heart disease — The intervention uses the brief and structured Sources of Meaning Card Method (SoMeCaM; www.somecam.org), which has been adapted for use in cardiac rehabilitation. It explores personal sources of meaning in a conversation with one patient in a 1-hour session. It comprises 26 cards each including statements on a particular source of meaning. The patient prioritizes the cards, reflects on them, and identifies possibilities for change.
  The conversation is facilitated by a professional (trained master students in psychology) and followed up with a phone call approximately 4 weeks after the conversation.
  Arms: a) Individual intervention format
Other: Group based session on Sources of Meaning in life with heart disease — The intervention is based on the brief and structured Sources of Meaning Card Method (SoMeCaM; www.somecam.org), which has been adapted for use in groups in a cardiac rehabilitation context. The method uses 26 cards, each representing a specific source of meaning. Approximately 6-10 participants are guided through a process of individually prioritizing the cards, reflecting on them and identifying potential areas for change or development in smaller groups. The group-based format enables mutual sharing and support in reflection and change processes among patients.
  The workshop is facilitated by a professional (trained master students in psychology) and followed up with individual phone calls with all participants approximately 4 weeks after the conversation.
  Arms: c) Group based intervention format
Other: Dyadic Conversation on Sources of Meaning in Life with heart disease — The intervention is based on the brief and structured Sources of Meaning Card Method (SoMeCaM; www.somecam.org), which has been adapted for use in dyads in a cardiac rehabilitation context. The method uses 26 cards, each representing a specific source of meaning. The dyadic format considers both the patient's and the relative's individual and shared sources of meaning in 1 session, which may enhance understanding for each other's sources of meaning and facilitate their joint daily life. They both prioritize the cards individually, reflect on them and identify possibilities for change through a talk-and-listen approach.
  The conversation is facilitated by a professional (trained master students in psychology) and followed up with a phone call approximately 4 weeks after the conversation.
  Arms: b) Dyadic (patient-relative) intervention format

SUMMARY:
Being diagnosed with heart disease can be a life-changing experience, often sparking existential questions and concerns about meaning in life. A lack of meaning in life has been found associated with increased emotional distress and decreased quality of life. Health professionals recognize that issues related to personal meaning in life are relevant but rarely address these aspects systematically in cardiac rehabilitation. This may be due to a lack of necessary tools.

The project evaluates a novel, brief and structured intervention that aims to strengthen the experience of meaningfulness and reduce or prevent emotional distress by addressing personal sources of meaning in life among patients attending cardiac rehabilitation and their relatives in Denmark. The intervention is based on the Sources of Meaning Card Method, a method developed by Peter la Cour and Tatjana Schnell to map and explore personal sources of meaning (www.somecam.org). For the current project, the method has been adapted for a cardiac rehabilitation context.

Three intervention formats are examined in a feasibility study in a municipal rehabilitation setting: 1) an individual format for patients in cardiac rehabilitation, 2) a dyadic format including a patient together with a relative, and 3) a group format for patients. Approximately 60 patients and 20 relatives are expected to participate. The study explores (a) participants' experience with and acceptability of the intervention formats; (b) changes in meaningfulness and emotional distress in a pre-post design; (c) recruitment and adherence rate, and (d) acceptability and practicality of the three formats among rehabilitation professionals.

ELIGIBILITY:
A.

Inclusion criteria, individual and group-based intervention formats:

* ≥18 years of age
* attending municipal cardiac rehabilitation
* proficiency in Danish

Exclusion criteria, individual and group-based intervention formats:

* severe psychiatric disorder
* severe cognitive impairment

B. Inclusion criteria, patients in dyadic intervention format

* as in A
* and having a relative who would like to participate

Inclusion criteria, relative in dyadic intervention format:

* ≥18 years of age
* relative to a patient attending municipal cardiac rehabilitation
* proficiency in Danish

Exclusion criteria, patient and relative dyadic intervention format

- as in A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Participants' experiences with the three intervention formats | Approximately 1 month post intervention
  Defined as the participants' experiences with their participation in one of the three intervention formats. Explored via focus groups and semi structured interviews.
Theoretical Framework of Acceptability (TFA) Questionnaire | 1 month post intervention
  Participants' acceptability of the intervention will be quantitatively assessed using the Theoretical Framework of Acceptability (TFA) Questionnaire. This scale evaluates the following seven constructs: affective attitude, burden, ethicality, opportunity costs, perceived effectiveness, self-efficacy, and intervention coherence.
  Each item is rated on a 5-point Likert scale ranging from 1 to 5. Higher scores indicate greater acceptability of the intervention across the measured domains.
Acceptability of the three intervention formats among participants | Approximately 1 month post intervention
  Acceptability will be explored qualitatively via focus groups and semi-structured interviews with participants enrolled in one of the three intervention formats
Changes in symptoms of depression | Baseline, 1 month post intervention and 3 months post intervention
  The Patient Health Questionnaire 9-item depression scale (PHQ-9) will be used to assess symptoms of depression in the past two weeks. Each item is scored 0 to 3. The severity score can range from 0 to 27, with higher scores indicating more severe symptoms.
Changes in symptoms of anxiety | Baseline, 1 month post intervention and 3 months post intervention
  The 7-item General Anxiety Disorder Scale (GAD-7) will be used to measure symptoms of anxiety in the past two weeks. Each item is scored 0 to 3, providing a 0 to 21 severity score, with higher scores indicating more severe symptoms.
Changes related to meaning in life | Baseline, 1 month post intervention and 3 months post intervention
  Changes in participants' self-reported experience of meaning in life will be assessed using two validated subscales from the Sources of Meaning and Meaning in Life Questionnaire: the Meaningfulness and Crisis of Meaning subscales.
  Each subscale consists of 5 items, scored on a Likert scale from 0 (Strongly disagree) to 5 (Strongly agree).
  For the Meaningfulness subscale, higher scores indicate a stronger sense of meaning in life.
  For the Crisis of Meaning subscale, higher scores indicate a stronger experience of life as empty, pointless and lacking of meaning.
Recruitment rate | From study start until recruitment ends (approximately 1 year)
  Recruitment rate is defined as the proportion of participants who consented to participate in the study, reported as a percentage over the recruitment period.
Intervention adherence | Through study completion, approximately 1 year
  The proportion of participants who completed the full intervention, defined as participation in the one-session Sources of Meaning conversation (individual, patient-relative, or group-based) and the follow-up phone call. Data will be recorded by the research team.
Study attrition (dropout rate) | Through study completion (approximately 15 months from study start)
  The proportion of participants who drop out from the study before completing all parts of the intervention, the 3 surveys and focus group and/or individual interview. Dropout will be assessed via administrative data.
Acceptability among rehabilitation professionals | After study enrollment (approximately 1 year from study start)
  Acceptability of the three intervention formats will be explored via focus groups with rehabilitation professionals involved in cardiac rehabilitation. The focus groups will address professionals' views on the interventions and perceived usefulness of the intervention in the municipal cardiac rehabilitation setting.
Practicality of the intervention formats among rehabilitation professionals | After study enrollment (approximately 1 year from study start)
  Defined as the rehabilitation professionals' evaluation of whether the intervention can be successfully used in practice (municipal cardiac rehabilitation). Including factors such as time, resources, and workflow compatibility. Explored via focus group with professionals in the municipal cardiac rehabilitation.
Intervention facilitators' experience with delivering the intervention | Through study completion (approximately 1 year from study start)
  Intervention facilitators will document their experience using semi-structured worksheets with field notes completed after each intervention session. These will capture reflections on feasibility, participant responsiveness, and challenges encountered in each step of the intervention.

SECONDARY OUTCOMES:
Changes in health-related quality of life | Baseline, 1 month post intervention and 3 months post intervention
  Explores changes in participants' self-reported health-related quality of life measured by EuroQol 5-Dimension 5-Level questionnaire (EQ-5D-5L).
  The EQ-5D-5L consists of 2 scales: the descriptive system (EQ-5D) and the EQ visual analogue scale (EQ VAS).
  EQ-5D measures the five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each with 5 levels from 'no problems', 'slight problems', 'moderate problems', 'severe problems' to 'extreme problems'.
  EQ VAS captures the participant's self-rated health on a vertical visual scale from 0-100 where 100 means: 'The best health you can imagine' and 0 means 'The worst health you can imagine'.
  Higher scores indicate better self-reported health-related quality of life.
Changes in awareness on sources of meaning in everyday life. | Baseline, 1 month post intervention and 3 months post intervention
  Changes in awareness on sources of meaning in everyday life will be explored using a purpose-designed self-report measure with 2 items covering awareness rated on a Likert scale ranging from 0 (Strongly disagree) to 5 (Strongly agree). Higher scores indicate greater awareness on sources of meaning in everyday life.
Changes in engagement in sources of meaning in everyday life | Baseline, 1 month post intervention and 3 months post intervention
  Changes in engagement in sources of meaning in everyday life will be explored using purpose-designed self-report measure with 3 items covering engagement rated on a Likert scale ranging from 0 (Strongly disagree) to 5 (Strongly agree). Higher scores indicate greater engagement on sources of meaning
Changes in mutual understanding (dyadic intervention arm) | Baseline, 1 month post intervention and 3 months post intervention
  Mutual understanding between patients and relatives in the dyadic intervention format will be assessed using the Understanding Subscale of the Perceived Partner Responsiveness Scale (PPRS) (Reis & Carmichael, 2006).
  The subscale consists of 5 items rated on a 9-point Likert scale ranging from 1 (Not at all true) to 9 (Very true). Higher scores indicate higher mutual understanding in the relationship to the other person.
Changes in relationship quality (dyadic intervention arm) | Baseline, 1 month post intervention and 3 months post intervention
  Relationship quality will be assessed using the Relationship Ladder, a single-item visual analogue scale in which participants rate their perceived relationship quality on a scale from 0 (Very poor) to 10 (Excellent).
  Higher scores indicate better perceived relationship quality.
Intervention costs | Through study completion (approximately 1 year post study start)
  To calculate intervention costs, information on time spent by intervention facilitators and other staff as well as material costs will be collected.
Reasons for dropout | At time of dropout (Up to 4 months post intervention)
  Reasons for participant dropout will be collected using a voluntary purpose-designed 3-item questionnaire at the time of dropout.
Engagement in intervention | 1 month post intervention
  Participant's engagement in the intervention is assessed through 2 purpose-designed questions: (1) 'Thought about the conversation at home' and (2) 'Used the reflection booklet at home'. Each question has an option to elaborate the answer qualitatively.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Center for Sundhed og Forebyggelse, Odense, Region Syddanmark
  - Sundhedskurser, Sundhedshus Vejle, Vejle, Region Syddanmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to Website of the Sources of Meaning Card Method. — https://somecam.org/